CLINICAL TRIAL: NCT07094542
Title: Temporo-masseteric Nerve Block in Post-wisdom Tooth Extraction Pain- a Randomized Study
Brief Title: Jaw Muscle Pain Post Wisdom Molar Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Gayathri Subramanian, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro2024001685
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Post Operative Pain; Impacted Third Molar Tooth; Muscle Pain
Keywords: Temporo-masseteric Nerve Block; Jaw muscle pain
MeSH Terms: conditions — Pain, Postoperative; Myalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant and investigators will be blinded to the treatment assignment- namely, the Temporo-masseteric Nerve Block using a placebo (sterile saline) or dental local anesthetic medication
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Active Comparator): Participants whose jaw muscle pain to palpation is <5 on Numerical Pain Rating Scale (NRS) the day after lower wisdom molar removal under sedation will be recommended post-operative pain management with a fixed interval dosing of ibuprofen 600 mg along with acetaminophen 325 mg taken every 6 hours for the first 72 hours post-procedure, after which they are encouraged to take prn dosing.
  Interventions: Drug: Oral Pain Medications only
- TMNB with Placebo (Active Comparator): Participants whose jaw muscle pain to palpation is 5 or higher on on Numerical Pain Rating Scale (NRS) the day after lower wisdom molar removal under sedation will be randomized to either placebo (sterile saline) or to the dental local anesthetic. The placebo will be delivered as the Temporo-masseteric Nerve Block injection. The randomization is blind to the participant and to the investigator administering the injection. The participants will be recommended post-operative pain management with a fixed interval dosing of ibuprofen 600 mg along with acetaminophen 325 mg taken every 6 hours for the first 72 hours post-procedure, after which they are encouraged to take prn dosing.
  Interventions: Drug: Temporo-masseteric Nerve Block Injection
- TMNB with dental local anesthetic (Experimental): Participants whose jaw muscle pain to palpation is 5 or higher on on Numerical Pain Rating Scale (NRS) the day after lower wisdom molar removal under sedation will be randomized to either placebo (sterile saline) or to the dental local anesthetic. The dental local anesthetic (2% lidocaine with 1:100,000 epinephrine) will be delivered as the Temporo-masseteric Nerve Block injection. The randomization is blind to the participant and to the investigator administering the injection. The participants will be recommended post-operative pain management with a fixed interval dosing of ibuprofen 600 mg along with acetaminophen 325 mg taken every 6 hours for the first 72 hours post-procedure, after which they are encouraged to take prn dosing.
  Interventions: Drug: Temporo-masseteric Nerve Block Injection

INTERVENTIONS:
Drug: Temporo-masseteric Nerve Block Injection — The TMNB injection/placebo will be administered by the Principal Investigator. The injection will only be delivered on Day 2 on the side/s of significant jaw muscle pain. Following disinfection of skin overlying the suprazygomatic injection site, a single carpule of 1.8 ml 2% lidocaine with 1:100,000 epinephrine will be delivered using a 25- or 27- gauge 30 mm needle). The injection site will be approximately a centimeter above the zygomatic arch, and a centimeter behind the palpable posterior border of the frontal process of the zygomatic bone. The needle will be directed at a 45-degree downward angle, directed medially along the coronal plane. At the depth of insertion of the needle, the local anesthetic/placebo will be delivered.
  Other Names: TMNB; Twin Block
  Arms: TMNB with Placebo; TMNB with dental local anesthetic
Drug: Oral Pain Medications only — For participants with jaw muscle pain to palpation <5 NRS score, no additional injection will be given. The participant will take the recommended pain medications as described.
  Arms: Control

SUMMARY:
The proposed design is a triple-blind, placebo-controlled randomized prospective phase II trial to assess the feasibility of employing the Temporo-masseteric Nerve Block (TMNB) injection to decrease jaw muscle pain, overall pain, improve mouth opening and minimize pain medication consumption. 80 participants undergoing lower third molar removal under sedation will be enrolled. Those who develop significant jaw muscle pain on the following day will be randomized to receive either the TMNB injection or a placebo. Daily ecological momentary assessments (EMAs) will be collected reflecting elements of patient experience for all participants. On Day 8, participants return for an end-of-study evaluation and return their unused pain medications. Up to 40 participants who are randomized to receive TMNB/placebo will be recruited to participate in a qualitative interview regarding their experience.

DETAILED DESCRIPTION:
The study is designed as a parallel, blinded, randomized phase II pilot study to assess the ability of the Temporo-masseteric Nerve Block (TMNB) injection to reduce post-operative pain in patients who undergo removal of lower third molar/s under sedation. It is not known how often and in whom jaw muscle pain significantly contributes to post-operative pain, limitation in mouth opening, and function. and develop significant jaw muscle pain. Hence the study is designed to assess the development of such jaw muscle pain before testing the placebo-controlled TMNB intervention. Accordingly, 80 subjects who undergo lower third molar extractions under intravenous sedation are randomized to receive either the TMNB (standard-of-care local anesthetic, 1.8 ml 2% lidocaine with 1:100,000 epinephrine), or a placebo (TMNB injection technique, but with 1.8 ml of sterile isotonic saline instead) the day following their extraction/s should they report significant pain (≥5 on a scale of pain rating from 0 to 10) when the jaw muscles are 'palpated' or examined with firm finger pressure. The assessment will be repeated 15 minutes after the injection. On the other hand, those who report less pain (<5) to jaw muscle palpation will not receive any injection. The participant, TMNB administrator and the evaluator will be blinded from randomization assignment. All participants will fill out daily remote surveys administered through REDCap® that will assess peak NRS pain score for the previous 24 hours, limitation in mouth opening and function, oral health related quality of life, pain medication consumption, and adverse effects from pain medications. Patient responses will be collected remotely and will include patient-uploaded cropped selfies of spontaneous mouth-opening with a disposable millimeter ruler (Orastretch®) propped between the upper and lower incisors.

It is anticipated that approximately 50% of patients will develop significant jaw muscle pain following the procedure. Hence, of the 80 participants, 40 are anticipated to be eligible for randomization, with 20 participants receiving the placebo or the TMNB injection, respectively.

Participants will return for an in-person assessment on Day 8, will return unused medications and will get an opportunity to participate in a qualitative interview to interrogate their experience receiving the injection (those randomized to TMNB/placebo), and their recovery experience. The duration of participation is a week from undergoing the procedure.

ELIGIBILITY:
Inclusion Criteria:

All patients recommended extraction/s of at least 1 lower wisdom (third) molar that is partially/fully 'impacted' under intravenous sedation, are eligible to participate in this study so long as they

* are 18 years or older,
* are healthy,
* have no cognitive/intellectual disability,
* have no past/recent pain or reduced range of motion in their jaw joint/ muscle complex, no trauma or surgery in their jaw region.
* have an electronic device such as a smart phone or a tablet/ computer with internet connection.
* are willing to participate in the study and not be excluded by the following criteria below.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Compromised ability to guard their self-interest, for e.g., prisoners, children, pregnant women, patients with intellectual/cognitive disability are not enrolled in the study.
* Those patients who present with infection/inflammation involving the third molars slated for extractions, on the day of their procedure, may not take part in the study.
* Those who have had opioid pain medication/s in the past 3 months to address short term or long-standing pain, or those who are on long term prescription of anti-inflammatory pain medication, are unable to participate.
* Those with long standing painful limitation of movement of the jaw joint or muscles.
* Those patients who are allergic to/unable to tolerate either the dental local anesthetic or its components, opioids, acetaminophen or ibuprofen also may not take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Jaw Muscle Pain Reduction on palpation post-TMNB injections | Day 2 15 minutes post TMNB injection
  To assess the effect of TMNB injection on the Numerical Pain Rating Scale (NRS) corresponding to Jaw muscle pain-to-palpation reported by the participant, when assessed 15 minutes post-injection.

SECONDARY OUTCOMES:
Sustained Benefit from TMNB Injection- pain reduction | 24-, 48-, 72-, and 96- hours post-injection
  Comparison of peak NRS pain score, the highest pain level as perceived by the participant collected for the preceding 24 hours.
Sustained Benefit from TMNB Injection- mouth opening | 24-, 48-, 72-, and 96- hours post-injection
  Comparison of spontaneous maximum mouth opening, measured in millimeters
Opioid consumption to 'rescue' pain poorly responsive to recommended pain medication regimen | 8 Days
  Compare need for rescue opioid medication among the three groups

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers School of Dental Medicine, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Final results will be posted no later than 12 months after the trial's primary completion date and will include participant flow, demographic and baseline characteristics, outcomes and statistical analyses, adverse events, the protocol, statistical analysis plan and administrative information.
  The PI will share the individual non-identified subject data no later than acceptance for the publication's main findings from the final data analysis or 18 months after completion of the study, whichever is earlier. Data to be posted will include the study protocol, reference to study publication of primary outcome variable, the data set in both SAS and ASCII formats, data dictionary and study specific de-identification notes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified data will be released within 12 months of primary completion date.
Access Criteria: Upon written request to the PI, survey instruments or other materials developed for use during the clinical trial will be made electronically available to other researchers.

REFERENCES:
- [Background] Subramanian G, Quek SYP. The Temporo-Masseteric Nerve Block (TMNB) for Alleviating Acute Postextraction Masticatory Myalgia: A Case Series. Anesth Prog. 2025 Mar 12;72(1):37-42. doi: 10.2344/24-0001. PMID 40657832
- [Background] Subramanian G, Makhija D, Ananthan S, Stitik TP, Quek SYP. Safety, efficacy, and mechanism of action of the temporo-masseteric nerve block. J Oral Facial Pain Headache. 2024 Jun;38(2):68-73. doi: 10.22514/jofph.2024.014. Epub 2024 Jun 12. PMID 39801096
- [Background] Quek SYP, Gomes-Zagury J, Subramanian G. Twin Block in Myogenous Orofacial Pain: Applied Anatomy, Technique Update, and Safety. Anesth Prog. 2020 Jun 1;67(2):103-106. doi: 10.2344/anpr-67-01-03. PMID 32633773
- [Background] Kanti V, Ananthan S, Subramanian G, Quek SYP. Efficacy of the twin block, a peripheral nerve block for the management of chronic masticatory myofascial pain: A case series. Quintessence Int. 2017 Oct 6:725-729. doi: 10.3290/j.qi.a39094. Online ahead of print. PMID 28990015
- [Background] Ananthan S, Kanti V, Zagury JG, Quek SYP, Benoliel R. The effect of the twin block compared with trigger point injections in patients with masticatory myofascial pain: a pilot study. Oral Surg Oral Med Oral Pathol Oral Radiol. 2020 Mar;129(3):222-228. doi: 10.1016/j.oooo.2019.09.014. Epub 2019 Oct 13. PMID 32009005